CLINICAL TRIAL: NCT03937752
Title: The Role of 3D Endoanal Ultrasound in Management of Anal Fistulas
Brief Title: 3D Endoanal Ultrasound and Anal Fistula
Acronym: UFU
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: Ultrasound study 2018/201
Record Dates: First submitted 2019-04-29; First posted 2019-05-06 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Anal Fistula
Keywords: anal fistula; fistula in ano; endoanal ultrasound; 3D ultrasound; 3D ultrasonography; endoanal ultrasonography; diagnostics
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Anal fistula: Patients with anal fistulas, no previous fistula procedures. Ultrasound investigation done as a part of surgical treatment, such as loose seton or fistulotomy.
  Interventions: Other: 3D endodanal ultrasound

INTERVENTIONS:
Other: 3D endodanal ultrasound — Endoanal ultrasound performed with two different transducers preoperatively during a fistula treatment procedure.
  Other Names: 3D endoanal ultrasonography

SUMMARY:
The study aims to evaluate the use of 3D endoanal ultrasound in preoperative management of anal fistula disease.

ELIGIBILITY:
Inclusion Criteria:

* anal fistula
* no previous fistula procedures

Exclusion Criteria:

* previous fistula procedures
* ano/rectovaginal fistula
* inflammatory bowel disease
* more than one internal openings

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with newly diagnosed anal fistula with no previous anal fistula procedures.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Fistula position | Day 1
  Dorsal? Ventral? Lateral - right or left?
Fistula level | Day 1
  Level I-IV (how much of the sphincter is affected?)
Fistula length | Day 1
  Shorter or longer than 3 cm?

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Aho Fält, MD, Principal Investigator — Region Skane
Locations (1):
- Pelvic Floor Centre, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Undecided